CLINICAL TRIAL: NCT07059013
Title: A Chatbot-based Program to Promote Well-being in Caregivers of Children With Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Wendy Zhang Wen, Assistant Professor, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: HMRFASDchatbot
Record Dates: First submitted 2025-04-30; First posted 2025-07-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot group (Experimental): The participants will be asked to communicate with the Chatbot.
  Interventions: Device: Chatbot
- Control group (No Intervention): One-page health information about ASD will be provided to the participants

INTERVENTIONS:
Device: Chatbot — The Chatbot will be designed using open-source conversational AI, such as GPT. The Chatbot will include three modules: individual strength, information, and Peer Networks.
  1. Individual Strength Include eight positive psychology exercises: positive introduction, personal strengths, using strengths, three good things, gratitude letter/visit, hope and optimism, active/constructive responding, and savoring.
  2. Information Include available healthcare services, parenting skills for children with ASD, the health information for ASD, the financial assistance provided by public and private funding, educational resources, and community resources.
  3. Peer Networks Participants can share their experiences about adapting after their child's diagnosis and read others' sharing.
  Arms: Chatbot group

SUMMARY:
Autism spectrum disorder (ASD) is characterized by varying degrees of disability and deviation in social communication, cognitive growth, and emotional expression, as well as the existence of constrained, repetitive patterns of behavior and interests and sensory processing issues. Caring for children with ASD can be a stressful and challenging life event for parents, potentially leading to a higher risk of mental health issues and other negative outcomes.

Poor mental health in these parents can be attributed to various factors, such as the perception of having little control over their child's behavior, concerns about the child's intellectual development and ability to acquire adaptive behaviors, the demands of caregiving and time management, worries about parent-child relationships, and uncertainty about the child's future.

The mental well-being of parents of children with ASD is essential in both clinical and research settings, as it can impact potential treatment results. Research has demonstrated that stress experienced by these parents can be linked to reduced participation in services and less favorable behavioral and developmental outcomes for their children in early intervention programs. The success of interventions mediated or delivered by parents is closely tied to their mental well-being, which affects both their involvement in treatments and adherence to them. Therefore, it is vital to focus on enhancing the mental health of parents when designing intervention children with ASD and their families.

Emerging evidence supports the use of Positive Psychotherapy (PPT). PPT was originally proposed by Seligman and colleagues and consists a series of evidenced-based positive psychological skills exercises aimed at fostering positive emotions, cognition, characteristics, and behaviors. PPT focuses on individuals' strengths and resources, distinguishing it from traditional psychotherapies. PPT is brief, requiring only a few sessions, Its instructions are straightforward and easy-to-follow, allowing for self-adminstration. Research has shown that PPT not only reduces depressive symptoms, stress and anxiety, but also places equal emphasis on enhancing well-being in individuals with major depression. Taken together, the investigators hypothesize that PPT can improve well-being, reduce stress, depressive symptoms, and enhance the quality of life in Chinese parents of children with ASD.

Digital health interventions, particularly Chatbots, have the potential to expand the reach and impact of positive psychology skills interventions for parents of children with ASD. There are several advantages to using Chatbots. First, Chatbots are perceived as accessible and can provide a structured set of content that simulates real-life conversations with a supportive friend. This is particularly important for parents of children with ASD who may lack social support. Second, access to the effective psychological interventions can be limited due to geographical barriers, lack of resources, or social stigma. Digital interventions, such as Chatbots, can help overcome these barriers by providing easy access to evidence-based psychological interventions. Chatbots can be available 24/7, can be personalized to individual needs, and can offer immediate feedback and support. Third, Chatbots can collect data on users' interactions, which can inform the improvement and adaptation of the intervention. The use of Chatbots to promote health conversations is an emerging field. A review of 12 studies suggested that no adverse events or harms were reported but there was a lack of studies assessing mental health outcomes. Hence, in this proposed study, the investigators will develop and test the first Chatbot to improve well-being in caregivers of children with ASD.

Aims： The objective is to evaluate and test the Chatbot-based program in promoting well-being in caregivers of children with ASD.

The secondary objectives are:

To test if the Chatbot-based program reduces perceived stress in caregivers of children with ASD; To test if the Chatbot-based program reduces depressive symptoms in caregivers of children with ASD; To test if the Chatbot-based program improves quality of life in caregivers of children with ASD; To test if the Chatbot-based program is feasible of children with ASD.

Methods: The randomised controlled trial with a mixed-method evaluation will be designed. A total of 130 caregivers of children with ASD will be randomly allocated into the control or intervention group. Participants will be randomly allocated to the Chatbot-based program and receive one-page information about ASD.

ELIGIBILITY:
Inclusion Criteria:

* caregivers providing long-term care for the children with a diagnosis of ASD from a qualified clinician, confirmed through the provision of documentation by the parents;
* caregivers of primary-school-age child (6-11 years old) (this age range is selected because social and communication interaction of children with ASD may be progressively more awkward in this age range when the social demands become more prominent);
* caregivers who are over 18 years old;
* caregivers who have the ability to communicate and read in Chinese;

Exclusion Criteria:

* Unwilling to complete the questionnaires at 3 time points;
* Diagnosis of severe psychiatric disorder (such as schizophrenia and severe bipolar disorder) or cognitive impairment;
* Participation of a similar psychological intervention within one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Well-being | Baseline, 3-month follow-up and 6-month follow-up
  Measured by the World Health Organization-5 Wellbeing Index (WHO-5) to evaluate vitality (being active and waking up fresh and rested), being interested in things, and having a pleasant attitude. Each item is scored using a 6-point Likert scale from at no time (0) to all of the time (5). The total score ranges from 0 to 25, with higher scores suggesting better self-perceived well-being.

SECONDARY OUTCOMES:
Depressive symptoms | Baseline, 3-month follow-up and 6-month follow-up
  Measured by the Patient Health Questionnaire-9 (PHQ-9), which evaluates the frequency of occurrence of main depressive symptoms over the past 2 weeks via a 4-point Likert scale from not at all (0) to nearly every day (3). The higher scores indicate more severe depressive symptoms.
Quality of life (QoL) | Baseline, 3-month follow-up and 6-month follow-up
  Measured by the Chinese version of Short-Form 12-item Survey-version 2 (SF-12v2), it consists of items that evaluate eight subscales pertaining to HRQOL, namely, role limitations due to physical restrictions (RP), physical functioning (PF), bodily pain (BP), general health compared with others (GH), vitality (VT), social functioning (SF), role limitations due to emotional issues (RE), and mental health (MH). The scores will be calculated by summing the relevant item responses and transforming the total to a 0-100 scale, following the standard scoring algorithm outlined in the Manual. Higher scores indicate better QoL.
Chatbot Feasibility (Quantitative outcome) | 3-month follow-up, 6-month follow-up
  Assessed by 2 items modified from the Feasibility of Intervention Measure. These 2 items will ask participants to evaluate that the Chatbot is implementable, and easy to use via a 5-point Likert scale from completely disagree (1) to completely agree (5). The total score ranges from 2 to 10, and higher scores indicate greater feasibility.
Parenting stress index | Baseline, 3-month follow-up and 6-month follow-up
  The Parenting Stress Index: Short Form (PSI-SF) consists of three subscales and a total stress score. The three subscales are parental distress (PD), parent-child dysfunctional interaction (PCDI) and difficult child (DC) score. The total stress score summarizes the three subscale scores (ranging from 36 to 180), and provides an overall indication of parenting stress. A Higher score indicates a higher level of parenting stress.

OTHER OUTCOMES:
Adverse events | through study completion, an average of 1 year
  Adverse events will be recorded during the program, which are defined as any unfavourable and unintended incidents that were not present initially or seem to have deteriorated from the baseline. The research team will evaluate the connection between these events and the study, while keeping track of their frequency and severity.
Chatbot feasibility (qualitative outcome) | 6-month follow-up
  The participants who attend the Chatbot-based program will be invited to this interview. Barriers and facilitators to participant adherence, and retention will be discussed in order to collect feedback. Interviews then specifically focused on discussing general needs in families of children with ASD and perspectives on potential feasibility, acceptability, facilitators, barriers, priority domains, and suggestions for the Chatbot.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Metropolitan University, Hong Kong, Hong Kong